CLINICAL TRIAL: NCT06714149
Title: Impacts of Nitrogen Deposition in the Natural Environment on Pollen Allergy in Belgium
Acronym: NITROPOL-BE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: prof. dr. Rik Schrijvers (Other)
Collaborators: Sciensano (Other Government); KU Leuven (Other); University of Namur (Other); UniversitÃ© Catholique de Louvain (Unknown)
Responsible Party: Sponsor-Investigator, prof. dr. Rik Schrijvers, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S65184; B2/212/P1/NITROPOL-BE (Other Grant/Funding Number: BELSPO)
Record Dates: First submitted 2024-11-20; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Pollen Allergy
Keywords: Nitrogen; Pollution; Pollen allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: A Cross-Sectional Paired Comparison Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergic subjects (Other): All subject with positive skin prick testing for grass and/or birch pollen are assigned to this group.
  Interventions: Diagnostic Test: Immunoreactivity testing
- Healthy controls (Other): Subjects with negative skin prick testing for grass and/or birch pollen are assigned to this group and used for as negative controls in our experiments.
  Interventions: Diagnostic Test: Immunoreactivity testing (negative control)

INTERVENTIONS:
Diagnostic Test: Immunoreactivity testing — Blood samples will be collected and used to determine the intensity of the allergenicity of the subject toward different types of pollen. This will be done by the detection of sIgE antibodies to the pollen extracts and basophil activation testing (BAT) with pollen extracts.
  Arms: Allergic subjects
Diagnostic Test: Immunoreactivity testing (negative control) — Blood samples will be collected and used to determine the background activity of our immunoreactivity tests. The investigators will use samples from negative controls to demonstrate that non-allergic individuals do not react to our assays, confirming that our pollen extracts have no background reactivity. This will be done by the detection of sIgE antibodies to the pollen extracts and basophil activation testing (BAT) with pollen extracts.
  Arms: Healthy controls

SUMMARY:
The investigators want to study the effect of environmental nitrogen enrichment on the allergy burden in pollen-sensitized subjects.

DETAILED DESCRIPTION:
The investigators want to study allergen-specific IgE reactivity from a cross-sectional sample of pollen-allergic patients (and negative controls) against environmental and experimental pollen samples. Following aspects will be compared:

* To study the basophil degranulation with different amounts of pollen on fresh patient-derived basophils, to determine the concentration of pollen needed to degranulate 5% (EC5), and 50% (EC50) of basophils.
* To study he overall intensity (quantitative), as well as IgE-mediated hyper- or hyporecognition of different fragments in the pollen samples (qualitative) in a subset of patients.
* To associate allergic rhinoconjunctivitis and food-pollen syndrome related symptoms with reactivity to different pollen samples.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test for grass and/or birch pollen

Exclusion Criteria:

* Desensitization therapy during the last two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Specific IgE reactivity (in-house developed) against environmental and experimental pollen samples | From time of inclusion to 12 months
  The investigators want to measure and compare sIgE values (kUA/L) towards different pollen samples.

SECONDARY OUTCOMES:
Basophil degranulation with different amounts of pollen on fresh patient-derived basophils. | From time of inclusion to 12 months
  The investigators want to measure and compare basophil degranulation with different pollen extracts on fresh patient-derived basophils. The investigators will use %CD63+ basophils as measure for basophil reactivity and sensitivity. The investigators will compare this between different pollen samples.
Overall intensity (quantitative) of IgE reactivity to pollen samples in a subset of patients. | From time of inclusion to 12 months
  The investigators will use an immunoblot to compare IgE mediated reactivity toward different pollen samples. Quantitatively, the investigators will compare band intensity (mean gray value) between different samples.
IgE-mediated hyper- or hyporecognition of different fragments in the pollen samples (qualitative) in a subset of patients. | From time of inclusion to 12 months
  The investigators will use an immunoblot to compare IgE mediated reactivity toward different pollen samples. Qualitatively, the investigators will compare presence of bands between samples.

OTHER OUTCOMES:
Association of allergic rhinoconjunctivitis symptoms with reactivity to different pollen samples (TNSS) | From time of inclusion to 12 months
  The Total Nasal Symptom Score (TNSS) is the sum of scores for each of nasal congestion, sneezing, nasal itching, and rhinorrhea at each time point, using a four point scale (0-3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 12.
Association of allergic rhinoconjunctivitis symptoms with reactivity to different pollen samples (VAS) | From time of inclusion to 12 months
  The rhinitis severity Visual analogue scale (VAS) is used to evaluate the overall severity of the rhinitis symptoms. The participant is asked to answer the several questions on: "How troublesome are your symptoms" on a 100mm VAS from 0 ('not troublesome') to 100 ('worst thinkable troublesome'). Based on their score on the VAS, the severity of rhinosinusitis can be divided into 3 categories as follows:
  Mild = VAS <20 mm Moderate = VAS 20-50 Severe = VAS >50
Association of allergic rhinoconjunctivitis symptoms with reactivity to different pollen samples (PFS) | From time of inclusion to 12 months
  Pollen-food syndrome (PFS) validated diagnostic questionnaire evaluates presence and severity of cross-reactivity. The diagnostic questionnaire and algorithm is a practical and robust tool, which enables rapid identification, and therefore management, of individuals with PFS who experience rhino-conjunctivitis symptoms in the birch pollen season. Evaluate association of cross-reactivity with reactivity to different pollen samples.
Association of allergic rhinoconjunctivitis symptoms with reactivity to different pollen samples (EQ-5D-5L) | From time of inclusion to 12 months
  Stress and well-being: evaluate impact on patients life - Quality of life (EuroQol 5 Dimensions, 5 Levels = EQ-5D-5L). Will be evaluated according to the standard guidelines. A worse rhinitis control and a worse asthma control are associated with higher EQ-5D-5L levels, particularly regarding pain/discomfort and activity impairment. Worse rhinitis control is associated with worse anxiety/depression, and poor asthma control with worse mobility.
  The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health status.
Association of allergic rhinoconjunctivitis symptoms with reactivity to different pollen samples (WPAI + CIQ: AS) | From time of inclusion to 12 months
  Allergy-Specific Work Productivity and Impairment (including CIQ = Classroom Impairment Questions) questionnaire (WPAI+CIQ: AS). Impaired work productivity has been associated with the severity of allergic rhinitis.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
  Scores:
  Multiply scores by 100 to express in percentages. Percent work time missed due to allergy: Q3/Q2 Percent impairment while working due to allergy: Q4/10 Percent overall work impairment due to allergy: (Q3/Q2)+[(1-(Q3/Q2))x(Q4/10)] Percent class time missed due to allergy: Q7/Q6 Percent impairment in the classroom due to allergy: Q8/10 Percent overall classroom impairment due to allergy: (Q7/Q6)+[(1-(Q7/Q6))x(Q8/10)] Percent activity impairment due to allergy: Q9/10

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verscheure P, Honnay O, Speybroeck N, Daelemans R, Bruffaerts N, Devleesschauwer B, Ceulemans T, Van Gerven L, Aerts R, Schrijvers R. Impact of environmental nitrogen pollution on pollen allergy: A scoping review. Sci Total Environ. 2023 Oct 1;893:164801. doi: 10.1016/j.scitotenv.2023.164801. Epub 2023 Jun 14. PMID 37321510
- [Background] Ceulemans T, Verscheure P, Shadouh C, Van Acker K, Devleesschauwer B, Linard C, Dendoncker N, Speybroeck N, Bruffaerts N, Honnay O, Schrijvers R, Aerts R. Environmental degradation and the increasing burden of allergic disease: The need to determine the impact of nitrogen pollution. Front Allergy. 2023 Feb 2;4:1063982. doi: 10.3389/falgy.2023.1063982. eCollection 2023. No abstract available. PMID 36819832